CLINICAL TRIAL: NCT05633875
Title: Multimodal Imaging Signatures of the Biological Mechanisms Underlying Neurodegeneration in Multiple Sclerosis: Long Term Predictive Value (IMAGIN-DEAL in MS)
Brief Title: Multimodal Imaging Signatures of the Biological Mechanisms Underlying Neurodegeneration in Multiple Sclerosis
Acronym: IMAGINDEALinMS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220766
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple sclerosis (MS); MRI; RRMS; long term predictive value; PET-MRI
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — Patients will undergo MRI without contrast agent

SUMMARY:
Multiple sclerosis (MS) is a chronic disease of the central nervous system characterised by multi-focal inflammatory and demyelinating lesions disseminated in the brain and in the spinal cord. Impressive advancements in the treatment of the autoimmune component of the disease have been achieved during the last decades, leading to a drastic reduction of white matter lesion accumulation and relapse rate along the disease course. However, the development of treatments effective for preventing or delaying the neurodegenerative component of the disease, that underly disability accrual and progression of the disease, remains a major challenge. The development of novel therapeutic strategies for neuroprotection that target all patients with MS is a priority objective for research in the next years. The critical steps towards identifying treatments that prevent neuro-axonal damage include a deep understanding of the mechanisms underlying neurodegeneration and the development of reliable biomarkers for assessing the efficacy of emerging drugs and for accelerating their translation to clinical use.

The team of Prof. Stankoff has pioneered an innovative imaging approach combining positron emission tomography and MRI, and succeeded in generating individual maps or key biological processes such as endogenous remyelination, neuroinflammation, or early damage preceding lesion formation. Using these approaches, it has been shown that these mechanisms were influencing disability worsening over the disease course, but the investigators still lack long term longitudinal studies for the validation of these advanced imaging metrics as prognosis markers. Recently, preliminary results have also suggested that a multimodal combination of advanced MRI sequences may have the potential to reproduce some PET results.

In this project the investigators propose to unravel the predictive value of individual maps of tremyelination, neuroinflammation, and early tissue damage, on long term disability worsening and to develop a novel imaging approach that aims to capture remyelination of lesions, ongoing inflammation invisible on T1 and T2 MRI sequences (subacute/chronic active lesions) and to predict short-term future disease activity (identify prelesional areas), from a single multimodal MRI acquisition in patients with MS.

DETAILED DESCRIPTION:
MS patient already included in previous studies using MRI and/or PET-MR (INFLASEP (NCT02305264), FLUMATEP (NCT01651520) or SHADOWTEP) will be proposed a long-term follow up study.

Participants will undergo :

* a full neurological examination including EDSS
* medical history and comorbidities (including smoking)
* concomitant and MS treatments
* neuropsychological testing
* Blood sample for serum biobanking
* multimodal MRI

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis Patient already enrolled in one of those 3 protocols since 8 years or more: INFLASEP, FLUMATEP 1-2 or SHADOWTEP
* Adult patient
* Affiliation to a social security scheme or beneficiary of such a scheme (Except "Aide Médicale d'Etat")
* Consent obtained

Exclusion Criteria:

* Any reasons, which does not allow to perform MRI, including claustrophobia, the implant of a pace maker or the presence of an intra-ocular foreign body (a contra- indication questionnaire will be filled in beforehand)
* Pregnancy, breast-feeding, lack of efficient contraception
* Current symptoms of severe or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary or cardiac disease, or any other chronic neurological diseases
* Unwillingness to be informed in case of abnormal MRI (with a significant medical anomaly)
* Enrolment in another interventional study protocol for the duration of his or her participation without physician's agreement
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subjects with Multiple Sclerosis will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
EDSS (Expanded Disability Status Scale) score | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression of neurological disability between the first inclusion in FLUMATEP, INFLASEP or SHADOWTEP study, and the inclusion in the current study. Scale: min=0 ;max=10

SECONDARY OUTCOMES:
MSFC (Component of the Multiple Sclerosis Functional Score) score for neurological disability: 9-Hole Peg Test (9HPG) | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=300
SDMT(Symbol Digit Modalities Test) for speed processing | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=110
T25FW (Timed 25 Foot Walk test) | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=180
MSFC (component of the Multiple Sclerosis Functional Score) score for neurological disability: PASAT (Paced Auditory Serial Addition Test) 3 sec for speed processing. Scale: min=0 ;max=60 | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS)
10/36 Spatial Recall tests | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=30
RL/RI-16 memory test | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=100
Backward and forward verbal digit span test | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=48
Stroop test | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=100
Deno 80 test | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS). Scale: min=0 ;max=80
White matter lesion load on MRI | Inclusion
  predictive value of imaging signatures (chronic active lesions, remyelination and prelesion areas) on the progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS)
Whole brain, white matter, deep grey matter and cortical atrophy on MRI | Inclusion
  Progression between baseline (inclusion in a first study: FLUMATEP, INFLASEP or SHADOWTEP) and follow up (IMAGIN-DEAL in MS)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Stankoff, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Olivier Colliot, Mr, Study Director — ARAMIS team (ICM) - Hospital Pitié-Salpêtrière
Locations (1):
- CIC Neurosciences, Paris, France